CLINICAL TRIAL: NCT02703740
Title: Long Term Safety and Efficacy Assessment of Hyaluronic Acid Dermal Filler With for the Treatment of Nasolabial Folds
Acronym: ECLAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Genévrier (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15F/IALE01
Record Dates: First submitted 2016-01-18; First posted 2016-03-09 (Estimated); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Aesthetics

ARMS (2):
- HA 20 mg/mL (Experimental)
  Interventions: Device: Hyaluronic acid dermal filler with lidocaine 0.3%
- HA 24 mg/mL (Experimental)
  Interventions: Device: Hyaluronic acid dermal filler with lidocaine 0.3%

INTERVENTIONS:
Device: Hyaluronic acid dermal filler with lidocaine 0.3% — injection in labial fold of a dermal filler

SUMMARY:
This study evaluates the injection of a hyaluronic acid dermal filler with lidocaine 0.3% in the treatment of nasolabial folds (NLF). Each patient will receive 1 concentration in a NLF (20 mg/mL) and an other concentration in the other NLF (24 mg/mL).

DETAILED DESCRIPTION:
Interventional, monocentric, double blind, randomised study Evaluation of safety the 1st month (primary criteria) and until 12 month Evaluation of performance at baseline, month 3, month 6, month 9 and month 12 : WSRS (wrinkle scale), profilometry (image measuring wrinkle depth and area), GAIS : satisfaction scale

ELIGIBILITY:
Inclusion Criteria:

* Is at least 19 years of age.
* Has Fitzpatrick Skin Type IV, V, or VI.
* Has a WSRS score > or = to 3 for both NLF
* Understands and accepts the obligation not to receive any other procedures or treatments in the nasolabial fold for 6 months

Exclusion Criteria:

Has keloid formation, or hypertrophic scarring or dyschromic scaring. Has hypersensitivity to hyaluronic acid, Chlorhexidine lidocaine or local anaesthetic drugs

* Has a known bleeding disorder or is receiving drug therapy that could increase the risk of bleeding.
* Has nasolabial folds that are too severe to be corrected in one treatment session.
* Has received any dermal filler or other injections, grafting or surgery in either nasolabial fold during the last year.
* Is pregnant, lactating, or not using acceptable contraception.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2017-02-03 (Actual); Study Completion 2017-02-03 (Actual)

PRIMARY OUTCOMES:
Number and description of adverse events that are related to treatment | 1 month

SECONDARY OUTCOMES:
Number and description of adverse events that are related to treatment | 72h/3 months/6 Months/9 months/12 months
Treatment efficacy assessed by WSRS | 1/3/6/9/12 months
  WSRS (wrinkle severity rating scale) : a 5-point validated scale ranging from 1 (absent) to 5 (extreme).

CONTACTS AND LOCATIONS:
Locations (1):
- CREABIO, Lyon, France